CLINICAL TRIAL: NCT02000154
Title: Phase I Clinical Trial of SyB L-1101 in Patients With Myelodysplastic Syndrome - Extension Study
Brief Title: Long Term Safety Study of SyB L-1101 in Patients With Recurrent/Relapsed or Refractory Myelodysplastic Syndrome (MDS) - Extension Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012001
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (1):
- SyB L-1101 (Experimental)
  Interventions: Drug: SyB L-1101

INTERVENTIONS:
Drug: SyB L-1101 — SyB L-1101 (rigosertib sodium) will be administered intravenously 72 continuous hours (3 days), followed by 25-day observation period. The treatment period of 28 days (3 days of administration + 25 days of observation) constitutes 1 cycle. The dose at cycle 8 in the study 2011005 will be the dose (if needed, the dose can be reduced) at the first cycle in this study (cycle 9). From cycle 10 on, the dose of SyB L-1101 will be reduced, delayed, or discontinued according to adverse events and results of observation at the previous cycle.

SUMMARY:
This is an extension study study to investigate long term safety of SyB L-1101 when administered intravenously every 4 weeks to the patients who have completed 8 cycles in the study 2011005 whose purpose is to investigate tolerability of SyB L-1101 when administered intravenously in patients with recurrent/relapsed or refractory myelodysplastic syndrome. Antitumor effects will also be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following conditions listed below.

1. Patients enrolled in the study 2011005 of SyB L-1101 in Patients With Myelodysplastic Syndrome.
2. Patients who was not judged as disease progression* nor progressive disease/relapsed** at the end of the cycle 8 in the study 2011005. * hematologic remission according to IWG 2006 criteria ** hematologic improvement according to IWG 2006 criteria
3. Patients who met the continuation criteria*** after Cycle 8 week 2 (Day 15±3) in the study 2011005.***defined in the study 2011005 protocol
4. Patients who can be expected to survive at least three months or longer.
5. Patients who have score of 0 to 2 in Eastern Cooperative Oncology Grou (ECOG) Performance Status (P.S.).
6. Patients with adequate function in major organs (heart, lungs, liver, kidneys, etc.).

   * Aspartate aminotransferase (AST): no more than 3.0 times the upper boundary of the reference range at each institution
   * Alanine aminotransferase (ALT): no more than 3.0 times the upper boundary of the reference range at each institution
   * Total bilirubin: no more than 1.5 times the upper boundary of the reference range at each institution
   * Serum creatinine: no more than 1.5 times the upper boundary of the reference range at each institution
   * ECG: no abnormal findings requiring treatment
   * Echocardiography: no abnormal findings requiring treatment
7. Patients who personally signed an informed consent document for participation in this study.

Exclusion Criteria:

Patients who satisfy any of the following conditions will not be enrolled in the study.

1. Patients with anemia (haemolytic anaemia, gastrointestinal haemorrhage, etc.) caused by factors other than MDS.
2. Patients with obvious infectious diseases (including viral infections).
3. Patients with serious complications (liver failure, renal failure, etc.).
4. Patients with a complication of serious heart disease (myocardial infarction, ischemic heart disease, etc.)
5. Patients with a serious gastrointestinal condition (severe or significant nausea/vomiting, diarrhea, etc.)
6. Patients with serious bleeding tendencies (disseminated intravascular coagulation (DIC), internal hemorrhage, etc.).
7. Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <130 milliequivalent/L).
8. Patients with an addiction to a legal or illegal drug, or with alcohol dependency.
9. Patients who are nursing, pregnant or may become pregnant.
10. Patients who have not consented to the following contraceptive measures. Patients will avoid sexual intercourse with sexual partners or should use the following contraceptive methods in these time periods: for male patients during the administration period of the trial and for six months after the end of administration; female patients during the administration period of the trial, and until a second menstrual period is confirmed after the end of administration (or in the case of female patients with no menstrual period, for two months after the end of administration). (1) Male patients:The patient will always use a condom. For effective contraception, it is recommended that the female partner also use the contraceptive methods for female patients. (2) Female patients: Female patients who may become pregnant should use one or more types of the following contraceptive methods. In addition, the male partner will always use a condom.

    * Oral contraceptive (birth control pills)
    * Intrauterine device (IUD)
    * Tubal ligation
11. Other patients judged to be unsuitable by an investigator or sub-investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Goto, Study Director — SymBio Pharmaceuticals
Locations (9):
- Japan (9):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kagoshima, Kagoshima-ken
  - Research site, Isesaki, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Sendai, Miyagi
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Kawagoe, Saitama
  - Research Site, Tokyo, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- SyB L-1101: SyB L-1101 （rigosertib sodium for intravenous formulation）:
  A 72-hour continuous intravenous dosing of SyB L-1101 4 weeks apart were administered to patients who had no disease progression of the primary disease at the end of the eighth cycle of Study 2011005, as well as those who gave consent to the continuous administration. The dose of SyB L-1101 in the ninth cycle was to be the same as that of the eighth cycle of Study 2011005 (if a dose reduction in the next cycle applied to a patient, SyB L-1101 was administered to the patient at the reduced dose).
Period: Overall Study
Arm/Group | SyB L-1101
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SyB L-1101
Number analyzed (Participants) | 1
Age, Customized [Number; unit: participants]
  60-69 years | 0
  70-79 years | 1
  80- years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Total number affected by any adverse events (details are presented in adverse event section)
Time Frame: Up to 20 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Disease Response Assessment
Description: Disease progression
  According to the International Working Group 2006 response criteria for Myelodysplastic Syndrome, "disease progression" is defined as no evidence of complete remission (CR), partial remission, marrow CR, stable disease, or failure, and as meeting one of the following conditions.
  1. when pretreatment percentage of bone marrow blasts < 5%: ≥ 50% increase to > 5%.
  2. when pretreatment percentage of bone marrow blasts 5 to 10%: ≥ 50% increase to > 10%.
  3. when pretreatment percentage of bone marrow blasts 10 to 20%: ≥ 50% increase to > 20%.
  4. when pretreatment percentage of bone marrow blasts 20 to 30%: ≥ 50% increase to > 30%.
  5. other: at least one of the following: decrease to ≤ 50% of neutrophil or platelet count at maximum response, ≥ 2 g/dL decrease in Hgb or transfusion dependence (in the absence of other factors, such as infection, gastrointestinal bleeding, or hemolysis).
Time Frame: Up to 20 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101
Number analyzed (Participants) | 1
participants | 1

3. Secondary Outcome: Serious Adverse Events
Description: Total number affected any serious adverse events
Time Frame: Up to 20 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101
Number analyzed (Participants) | 1
participants | 0

4. Secondary Outcome: Hematologic Improvement
Description: NCA (not considered assessable)
  no evidence of hematologic improvement -erythroid, -platelet, -neutrophil, progressive disease, or relapse, defined in the International Working Group 2006 response criteria for myelodysplastic syndrome.
Time Frame: Up to 20 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101
Number analyzed (Participants) | 1
participants | 1

5. Secondary Outcome: Cytogenetic Response
Description: NCA (not considered assessable)
  no evidence of cytogenetic response, defined in the International Working Group 2006 response criteria for myelodysplastic syndrome.
Time Frame: Up to 20 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-1101
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Arm/Group | SyB L-1101
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB L-1101 (N=1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No